CLINICAL TRIAL: NCT00343915
Title: Long-term Study of Immune Response Persistence of GSK Biologicals' 2-dose Thiomersal-free Engerix™-B and 3-dose Preservative-free Engerix™-B Vaccines in Subjects Aged 11-15 Yrs
Brief Title: Immuno & Safety Study of GSK Biologicals' Thio or Preservative Free Hepatitis B Vaccine in Subjects Aged 11-15 Yrs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 101695 Ext. Mth30; 101696 (Other: GSK); 101697 (Other: GSK); 101698 (Other: GSK); 2015-001531-20 (EudraCT Number); NCT00787228 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2006-06-23 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis B
Keywords: Persistence; Hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- 2-Dose Engerix (Experimental): subjects received 2 doses of adult (thiomersal-free) HBV formulation, one at 0 and 6 months, respectively and placebo (physiological saline) at 1 month.
  Interventions: Biological: Engerix™-B (thiomersal-free) 20µg; Biological: placebo
- 3-Dose Engerix (Active Comparator): subjects received 3 doses of paediatric (preservative-free) HBV formulation one at 0, 1 and 6 months, respectively.
  Interventions: Biological: 10 μg Engerix™-B (preservative-free)

INTERVENTIONS:
Biological: Engerix™-B (thiomersal-free) 20µg — In the primary study: 2 deep intramuscular injections (Months 0, & 6)
  Arms: 2-Dose Engerix
Biological: 10 μg Engerix™-B (preservative-free) — In the primary study: 3 deep intramuscular injections (months 0, 1 & 6)
  Arms: 3-Dose Engerix
Biological: placebo — In the primary study: 1 deep intramuscular injection (month 1)
  Arms: 2-Dose Engerix

SUMMARY:
To evaluate the persistence of antibodies against hepatitis B at 30, 42, 54 and 66 months after the first dose of the hepatitis B primary vaccination course.

Subjects were aged 11 to 15 years at the time of the primary vaccination course.

At the time of enrollment in the present long-term follow-up study subjects were aged 13 to 18 years.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
All subjects who participated in the primary study, in which they received either 2 or 3 doses of GSK Biologicals hepatitis B vaccine, and who consented to participate in the long-term follow-up at Month 42 were contacted by the investigators.

No additional subjects will be recruited during this long-term follow-up study and no vaccine will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have participated in primary study HBV-280
* Written informed consent will be obtained from each subject and/ or parent or guardian of the subject before the blood-sampling visit of each year

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 267 (Actual)
Dates: Start 2004-04-21 (Actual); Primary Completion 2008-01-10 (Actual); Study Completion 2008-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Sydney, New South Wales, Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Wilrijk
- GSK Investigational Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Heron L, Selnikova O, Moiseieva A, Van Damme P, van der Wielen M, Levie K, Hoet B, Stoffel M. Immunogenicity, reactogenicity and safety of two-dose versus three-dose (standard care) hepatitis B immunisation of healthy adolescents aged 11-15 years: a randomised controlled trial. Vaccine. 2007 Apr 12;25(15):2817-22. doi: 10.1016/j.vaccine.2006.12.021. Epub 2006 Dec 29. PMID 17276552
- [Background] Heron LG, Chant KG, Jalaludin BB. A novel hepatitis B vaccination regimen for adolescents: two doses 12 months apart. Vaccine. 2002 Oct 4;20(29-30):3472-6. doi: 10.1016/s0264-410x(02)00346-8. PMID 12297392
- [Background] Van Damme P, Moiseeva A, Marichev I, Kervyn AD, Booy R, Kuriyakose S, Brockway A, Ng SP, Leyssen M, Jacquet JM. Five years follow-up following two or three doses of a hepatitis B vaccine in adolescents aged 11-15 years: a randomised controlled study. BMC Infect Dis. 2010 Dec 20;10:357. doi: 10.1186/1471-2334-10-357. PMID 21171982
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 101695 Ext. Mth30 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101695 Ext. Mth30 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101695 Ext. Mth30 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101695 Ext. Mth30 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 101695 (Ext HBV-280 M30) are summarised with studies 103860/280 (HBV-280), 101696 (Ext HBV-280 M42), 101697 (Ext HBV-280 M54) and 101698
- Available data/document: Dataset Specification: 101695 Ext. Mth30 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects who participated in the primary vaccination study, in which they received either 2 or 3 doses of GSK Biologicals hepatitis B vaccine, and who consented to participate in the long-term follow-up were contacted by the investigators. No additional subjects were recruited during this long-term follow-up study.
Period: Primary Study
Arm/Group | 2-dose Engerix | 3-dose Engerix
Started | 258 | 126
Completed | 254 | 123
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Other | 1 | 0
Period: Month 30 Follow-up
Arm/Group | 2-dose Engerix | 3-dose Engerix
Started | 179 (Subjects, previously vaccinated, that returned for the Month 30 follow-up.) | 88
Completed | 179 | 88
Not Completed | 0 | 0
Period: Month 42 Follow-up
Arm/Group | 2-dose Engerix | 3-dose Engerix
Started | 174 (Subjects, previously vaccinated, that returned for the Month 42 follow-up.) | 84
Completed | 174 | 84
Not Completed | 0 | 0
Period: Month 54 Follow-up
Arm/Group | 2-dose Engerix | 3-dose Engerix
Started | 166 (Subjects, previously vaccinated, that returned for the Month 54 follow-up.) | 79
Completed | 166 | 79
Not Completed | 0 | 0
Period: Month 66 Follow-up
Arm/Group | 2-dose Engerix | 3-dose Engerix
Started | 158 (Subjects, previously vaccinated, that returned for the Month 66 follow-up.) | 76
Completed | 158 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-dose Engerix | 3-dose Engerix | Total
Number analyzed (Participants) | 258 | 126 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (1.23) | 12.7 (1.32) | 12.8 (1.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 61 | 193
  Male | 126 | 65 | 191

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected for Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody.
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Time Frame: At Month 7
Population: The ATP cohort for immunogenicity included all evaluable subjects who had post-vaccination immunogenicity results and who complied with the protocol, including the time schedule for vaccination and blood sample draw.
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 241 | 113
Subjects | 233 | 111

2. Primary Outcome: Number of Subjects Seroprotected for Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody.
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Time Frame: At Month 30, Month 42, Month 54 and Month 66
Population: Long Term According-to-Protocol cohort for immunogenicity, including all subjects who returned at the considered follow-up time point and who complied with the protocol.
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 166 | 80
Subjects
  Month 30 (N=140, 64) | 122 | 62
  Month 42 (N=166, 80) | 139 | 74
  Month 54 (N=147, 76) | 124 | 72
  Month 66 (N=132, 70) | 105 | 64

3. Primary Outcome: Antibody Titers Against Hepatitis-B Virus.
Description: Antibody titers were summarized by Geometric Mean Concentrations (GMCs) with their 95% CIs.
Time Frame: At Month 30, Month 42, Month 54 and Month 66
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 166 | 80
mIU/mL
  Month 30 (N=140, 64) | 229.0 [162.1 to 323.5] | 708.3 [409.6 to 1224.8]
  Month 42 (N=166, 80) | 159.7 [118.3 to 215.7] | 417.9 [267.3 to 653.6]
  Month 54 (N=147, 76) | 123.6 [92.7 to 165.0] | 277.6 [176.5 to 436.7]
  Month 66 (N=132, 70) | 82.1 [60.7 to 111.0] | 225.2 [142.6 to 355.9]

4. Secondary Outcome: Antibody Titers Against Hepatitis-B Virus.
Description: Antibody titers were summarized by Geometric Mean Concentrations (GMCs) with their 95% CIs.
Time Frame: At Months 1, 2, 6 and 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 241 | 113
mIU/mL
  Month 1 (N=240, 112) | 28.8 [16.8 to 49.2] | 28.7 [9.4 to 87.8]
  Month 2 (N=240, 113) | 17.6 [11.1 to 27.8] | 29.4 [21.6 to 40.1]
  Month 6 (N=239, 113) | 18.8 [14.7 to 24.1] | 90.0 [68.6 to 117.9]
  Month 7 (N=241, 113) | 2738.5 [2071.4 to 3620.5] | 7238.3 [5247.3 to 9984.7]

5. Secondary Outcome: Number of Subjects Seroprotected for Anti-HBs Antibody.
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Time Frame: At Months 1, 2 and 6
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 240 | 113
Subjects
  Month 1 (N=240, 112) | 31 | 8
  Month 2 (N=240, 113) | 27 | 63
  Month 6 (N=239, 113) | 63 | 99

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccination and overall
Population: The ATP cohort for safety included all evaluable subjects, who received at least one dose of study vaccine according to their random assignment, with sufficient data to perform safety analysis, who did not receive a vaccine not specified or forbidden in the protocol.
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 253 | 121
Subjects
  Any Pain; Dose 1 (N=253, 121) | 121 | 44
  Grade 3 Pain; Dose 1 (N=253, 121) | 6 | 3
  Any Redness; Dose 1 (N=253, 121) | 30 | 10
  Grade 3 Redness; Dose 1 (N=253, 121) | 0 | 1
  Any Swelling; Dose 1 (N=253, 121) | 18 | 8
  Grade 3 Swelling; Dose 1 (N=253, 121) | 2 | 2
  Any Pain; Dose 2 (N=252, 119) | 42 | 38
  Grade 3 Pain; Dose 2 (N=252, 119) | 3 | 2
  Any Redness; Dose 2 (N=252, 119) | 15 | 15
  Grade 3 Redness; Dose 2 (N=252, 119) | 1 | 0
  Any Swelling; Dose 2 (N=252, 119) | 8 | 5
  Grade 3 Swelling; Dose 2 (N=252, 119) | 1 | 0
  Any Pain; Dose 3 (N=250, 118) | 106 | 35
  Grade 3 Pain; Dose 3 (N=250, 118) | 4 | 1
  Any Redness; Dose 3 (N=250, 118) | 29 | 11
  Grade 3 Redness; Dose 3 (N=250, 118) | 0 | 0
  Any Swelling; Dose 3 (N=250, 118) | 14 | 6
  Grade 3 Swelling; Dose 3 (N=250, 118) | 0 | 0
  Any Pain; Across Doses (N=253, 121) | 155 | 74
  Grade 3 Pain; Across Doses (N=253, 121) | 8 | 6
  Any Redness; Across Doses (N=253, 121) | 50 | 28
  Grade 3 Redness; Across Doses (N=253, 121) | 0 | 1
  Any Swelling; Across Doses (N=253, 121) | 27 | 15
  Grade 3 Swelling; Across Doses (N=253, 121) | 2 | 2

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache, and fever. Any was defined as incidence of the specified symptoms regardless of intensity or relationship to study vaccine. Gastrointestinal symptoms included nausea, vomiting, diarrhea and abdominal pain. Grade 3 fever was defined as fever (axillary temperature) > 38.5°C. Grade 3 symptoms were defined as symptoms which prevented normal everyday activities. Related = general symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccination and overall
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 253 | 121
Subjects
  Any Fatigue; Dose 1 (N=253, 121) | 50 | 26
  Grade 3 Fatigue; Dose 1 (N=253, 121) | 1 | 1
  Related Fatigue; Dose 1 (N=253, 121) | 29 | 16
  Any Gastrointestinal; Dose 1 (N=253, 121) | 26 | 4
  Grade 3 Gastrointestinal; Dose 1 (N=253, 121) | 3 | 0
  Related Gastrointestinal; Dose 1 (N=253, 121) | 11 | 3
  Any Headache; Dose 1 (N=253, 121) | 57 | 29
  Grade 3 Headache; Dose 1 (N=253, 121) | 0 | 1
  Related Headache; Dose 1 (N=253, 121) | 33 | 15
  Any Temperature; Dose 1 (N=253, 121) | 4 | 2
  Grade 3 Temperature; Dose 1 (N=253, 121) | 0 | 0
  Related Temperature; Dose 1 (N=253, 121) | 3 | 2
  Any Fatigue; Dose 2 (N=252, 119) | 37 | 18
  Grade 3 Fatigue; Dose 2 (N=252, 119) | 2 | 0
  Related Fatigue; Dose 2 (N=252, 119) | 23 | 13
  Any Gastrointestinal; Dose 2 (N=252, 119) | 20 | 7
  Grade 3 Gastrointestinal; Dose 2 (N=252, 119) | 0 | 0
  Related Gastrointestinal; Dose 2 (N=252, 119) | 7 | 5
  Any Headache; Dose 2 (N=252, 119) | 40 | 21
  Grade 3 Headache; Dose 2 (N=252, 119) | 0 | 0
  Related Headache; Dose 2 (N=252, 119) | 24 | 11
  Any Temperature; Dose 2 (N=252, 119) | 5 | 5
  Grade 3 Temperature; Dose 2 (N=252, 119) | 1 | 0
  Related Temperature; Dose 2 (N=252, 119) | 5 | 4
  Any Fatigue; Dose 3 (N=250, 118) | 49 | 20
  Grade 3 Fatigue; Dose 3 (N=250, 118) | 3 | 2
  Related Fatigue; Dose 3 (N=250, 118) | 30 | 8
  Any Gastrointestinal; Dose 3 (N=250, 118) | 17 | 14
  Grade 3 Gastrointestinal; Dose 3 (N=250, 118) | 3 | 2
  Related Gastrointestinal; Dose 3 (N=250, 118) | 6 | 6
  Any Headache; Dose 3 (N=250, 118) | 36 | 20
  Grade 3 Headache; Dose 3 (N=250, 118) | 1 | 1
  Related Headache; Dose 3 (N=250, 118) | 22 | 12
  Any Temperature; Dose 3 (N=250, 118) | 13 | 9
  Grade 3 Temperature; Dose 3 (N=250, 118) | 1 | 0
  Related Temperature; Dose 3 (N=250, 118) | 7 | 5
  Any Fatigue; Across Doses (N=253, 121) | 77 | 46
  Grade 3 Fatigue; Across Doses (N=253, 121) | 4 | 3
  Related Fatigue; Across Doses (N=253, 121) | 51 | 30
  Any Gastrointestinal; Across Doses (N=253, 121) | 36 | 21
  Grade 3 Gastrointestinal; Across Doses (N=253,121) | 6 | 2
  Related Gastrointestinal; Across Doses (N=253,121) | 17 | 14
  Any Headache; Across Doses (N=253, 121) | 78 | 46
  Grade 3 Headache; Across Doses (N=253, 121) | 1 | 2
  Related Headache; Across Doses (N=253, 121) | 49 | 30
  Any Temperature; Across Doses (N=253, 121) | 17 | 14
  Grade 3 Temperature; Across Doses (N=253, 121) | 1 | 0
  Related Temperature; Across Doses (N=253, 121) | 10 | 10

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Event (AE).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day (Day 0-30) follow-up period after each vaccination and overall
Population: Total Cohort included all enrolled (i.e. randomized or vaccinated) subjects who received at least one vaccine dose and for whom data were available. No information regarding AEs was available for 1 subject in each group
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 257 | 125
Subjects
  any AE(s) | 112 | 54
  grade 3 AE(s) | 31 | 15
  related AE(s) | 9 | 1

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Month 0 to Month 66)
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 257 | 125
Subjects | 4 | 1

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: erious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: At Month 30, Month 42, Month 54 & Month 66
Population: LT total cohort included all subjects who were included in the total cohort in the primary study and returned at the considered follow-up time point.
Measure: Number; unit: Participants
Arm/Group | 2-dose Engerix | 3-dose Engerix
Number analyzed (Participants) | 179 | 88
Participants
  Month 30 (N=179, 88) | 0 | 0
  Month 42 (N=174, 84) | 0 | 0
  Month 54 (N=166, 79) | 0 | 0
  Month 66 (N=158, 76) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events: during the entire study period (Month 0-66), Solicited local and general symptoms: During the 4-day (Days 0-3) post vaccination period and unsolicited adverse events: up to Month 7.Non-serious adverse events were not assessed during the long term follow-up period (Month 30-66). The total number of participants at risk is the number of participants with at least one documented dose.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | 2-dose Engerix | 3-dose Engerix
All-Cause Mortality (participants affected / at risk) | 0/257 | 0/125
Serious Adverse Events (participants affected / at risk) | 4/257 | 1/125
Other Adverse Events (participants affected / at risk) | 155/257 | 74/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2-dose Engerix (N=257) | 3-dose Engerix (N=125)
Injury (Injury, poisoning and procedural complications) | 1 | 1
Arthritis (Infections and infestations) | 1 | 0
Ileitis (Gastrointestinal disorders) | 1 | 0
Infection bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 2-dose Engerix (N=257) | 3-dose Engerix (N=125)
Pain; Dose 1 (General disorders) | 121/253 | 44/121
Redness; Dose 1 (General disorders) | 30/253 | 10/121
Swelling; Dose 1 (General disorders) | 18/253 | 8/121
Pain; Dose 2 (General disorders) | 42/252 | 38/119
Redness; Dose 2 (General disorders) | 15/252 | 15/119
Pain; Dose 3 (General disorders) | 106/250 | 35/118
Redness; Dose 3 (General disorders) | 29/250 | 11/118
Swelling; Dose 3 (General disorders) | 14/250 | 6/118
Pain; Across Doses (General disorders) | 155/253 | 74/121
Redness; Across Doses (General disorders) | 50/253 | 28/121
Swelling; Across Doses (General disorders) | 27/253 | 15/121
Fatigue; Dose 1 (General disorders) | 50/253 | 26/121
Gastrointestinal symptoms; Dose 1 (Gastrointestinal disorders) | 26/253 | 4/121
Headache; Dose 1 (Nervous system disorders) | 57/253 | 29/121
Fatigue; Dose 2 (General disorders) | 37/252 | 18/119
Gastrointestinal symptoms; Dose 2 (Gastrointestinal disorders) | 20/252 | 7/119
Headache; Dose 2 (Nervous system disorders) | 40/252 | 21/119
Fatigue; Dose 3 (General disorders) | 49/250 | 20/118
Gastrointestinal symptoms; Dose 3 (Gastrointestinal disorders) | 17/250 | 14/118
Fever; Dose 3 (General disorders) | 13/250 | 9/118
Fatigue; Across Doses (General disorders) | 77/253 | 46/121
Gastrointestinal symptoms; Across Doses (Gastrointestinal disorders) | 36/253 | 21/121
Headache; Across Doses (Nervous system disorders) | 78/253 | 46/121
Fever; Across Doses (General disorders) | 17/253 | 14/121
Upper respiratory tract infection (Infections and infestations) | 26 | 22
Headache (Nervous system disorders) | 28 | 10
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 15 | 5
Headache; Dose 3 (Nervous system disorders) | 36/250 | 20/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.